CLINICAL TRIAL: NCT07333183
Title: An Open-Label, Phase 2 Study Evaluating the Safety of Mosliciguat in Combination With Inhaled Treprostinil in Participants With Pulmonary Hypertension Associated With Interstitial Lung Disease
Brief Title: A Study of Mosliciguat in Combination With Inhaled Treprostinil in PH-ILD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmovant, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVT-2301-202
Record Dates: First submitted 2026-01-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease (ILD); Lung Diseases; Vascular Diseases; Cardiovascular Diseases; Fibrosis
Keywords: PH; ILD; 6 Minute Walk Test; mosliciguat
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial; Lung Diseases; Vascular Diseases; Cardiovascular Diseases; Fibrosis | interventions — Dry Powder Inhalers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Active Comparator: inhaled mosliciguat (Experimental): Participants will receive inhaled mosliciguat daily for 16 weeks
  Interventions: Drug: inhaled mosliciguat; Device: Dry Powder Inhaler
- Extension: inhaled mosliciguat (Experimental): After Week 16, all participants will continue to receive inhaled mosliciguat through an Extension period
  Interventions: Drug: inhaled mosliciguat; Device: Dry Powder Inhaler

INTERVENTIONS:
Drug: inhaled mosliciguat — Dose level 1, 2, or 3 for inhalation
Device: Dry Powder Inhaler — Dry powder inhaler for mosliciguat delivery

SUMMARY:
This is a Phase 2, open-label, multi-center clinical study to evaluate the safety and efficacy of inhaled mosliciguat in participants with pulmonary hypertension associated with interstitial lung disease (PH-ILD) on a background inhaled treprostinil.

DETAILED DESCRIPTION:
This study is an open-label study with an extension.

The study consists of 2 periods: an open label treatment period (16 weeks) and an extension (beyond 16 weeks).

Participants will receive mosliciguat in the 16-week treatment period.

All participants who complete the 16-week treatment period may continue to participate in the extension period where all participants will receive mosliciguat.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing and able to provide informed consent
* Participants on inhaled treprostinil
* Participants with diagnosis of Interstitial Lung Disease (ILD). Diagnosis will be confirmed by a high-resolution computerized tomography (HR-CT) scan showing diffuse parenchymal disease. Eligible diagnosed diseases include:

  1. Idiopathic interstitial pneumonia (IIP)
  2. Chronic hypersensitivity pneumonitis
  3. ILD associated with connective tissue disease (CTD) with a forced vital capacity (FVC) < 70% of predicted
* Confirmed pulmonary hypertension (PH) by right heart catheterization (RHC).
* Ability to perform 6MWD ≥100 meters.

Exclusion Criteria:

* Diagnosis of PH Group 1 (eg. pulmonary arterial hypertension), Group 2 (related to left-heart dysfunction), Group 4 (eg, chronic thromboembolic pulmonary hypertension), or Group 5 (eg, unclassified).
* Exacerbation of underlying lung disease within 28 days prior to randomization.
* Initiation of pulmonary rehabilitation within 28 days prior to randomization.
* Receiving >10 L/min of oxygen supplementation by any mode of delivery at rest at Baseline.
* History or intolerance to or lack of efficacy with mosliciguat or sGC stimulators or activators.
* Receipt of investigational, or experimental therapy within 42 days OR 5 half-lives prior to randomization.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of participant TEAEs, SAEs, and AEs leading to discontinuation | Baseline, Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Ubaldo Martin, MD, Study Director — Pulmovant, Inc.
Locations (1):
- Florida Lung, Asthma & Sleep Specialists/Clinical Research Specialists, LLC, Kissimmee, Florida, United States